CLINICAL TRIAL: NCT05136079
Title: Prophylactic LYMphatic Reconstruction (LYMbR) to Prevent Lymphedema
Brief Title: Prophylactic LYMphatic Reconstruction (LYMbR) to Prevent Lymphedema After Node Dissection for Cutaneous Malignancies
Acronym: LYMbR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alberta Health Services, Calgary (Other)
Collaborators: University of Calgary (Other); Tom Baker Cancer Centre (Other)
Responsible Party: Principal Investigator, Claire Temple-Oberle, Surgeon, Departments of Surgery and Oncology; Professor - University of Calgary, Alberta Health Services, Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PLVA-2021
Record Dates: First submitted 2021-11-02; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Lymphedema of Limb; Malignant Skin Neoplasm
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: A total of 40 study participants will be block (axilla, groin) randomized using 2 equal groups (control/intervention) of 20 participants each.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant: Participants will not be informed of their study arm allocation until they complete the study. Regardless of study arm, participants will be injected with the requisite blue dye to perform the LVA procedures, thereby providing no visible clue as to whether they are control or intervention participants. The exception will be in the case where a participant is diagnosed with lymphedema post-operatively but prior to their study participation completion and their healthcare management requires knowledge of surgical history.
  Radiologist: At 24 months each participant will undergo a radionuclide lymphoscintigraphy to assess the functioning of the lymphatic system. The radiologist reading the results will be blinded as to the participants' study allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic lymphaticovenous anastomosis (Experimental): Intervention participants will undergo prophylactic lymphaticovenous anastomosis as an addendum to axillary or ilioinguinal lymphadenectomy for treatment of cutaneous malignancy.
  Interventions: Procedure: Prophylactic lymphaticonvenous anastomosis
- Lymphadenectomy without lymphaticovenous anastomosis (No Intervention): Control participants will undergo axillary or ilioinguinal lymphadenectomy without lymphaticovenous anastomosis for treatment of cutaneous malignancy .

INTERVENTIONS:
Procedure: Prophylactic lymphaticonvenous anastomosis — Prophylactic lymphaticovenous anastomosis is an immediate prophylactic approach whereby the lymphaticovenous anastomosis is performed at the time of nodal dissection utilizing fluorescing indocynanine green (ICG) and an operating microscope.
  Arms: Prophylactic lymphaticovenous anastomosis

SUMMARY:
Background: Lymphedema following lymph node dissection is a chronic condition that can limit physical, occupational, and social participation, impact self-image, and result in financial burden. Studies have reported lymphedema incidence rates of 39% to 73% following node dissection.

Lymphaticovenous anastomosis (LVA) has been previously used to treat established lymphedema. More recently, with imaging capabilities guided by blue dye and indocyanine green dye, the possibility of prophylactic LVA has become feasible. A 2018 systematic review of 12 studies utilizing prophylactic LVA during lymphadenectomy indicated a 2/3 reduction in the risk of lymphedema. The literature yet lacks any phase III studies with stringent controls and long term follow-up.

Objectives: To assess (primary endpoint) the impact of prophylactic LVA on presence or absence of lymphedema post axillary or groin lymphadenectomy and participant quality of life. To assess (secondary endpoint) the incidence of complications related to nodal dissection.

Methods: This is a phase III RCT, block randomized for upper and lower extremities, recruiting adult patients planned for an axillary or groin node dissection as a result of cutaneous malignancy. Analysis of rates of lymphedema and quality of life reports will be done.

Significance: Lymphedema is a feared outcome of surgical cancer care. Its impact on patients' daily lives is profound. A reduction of incidence of this debilitating condition by 2/3 would have significant impact on numerous lives and could also reduce the health system resources needed for its management.

DETAILED DESCRIPTION:
Trial Objective: To ascertain the efficacy and impact of prophylactic lymphaticovenous anastomosis for prevention of lymphedema in cutaneous malignancy patients undergoing axillary or groin node dissection as part of cancer treatment. To determine quality of life impact, if any, for patients who receive this treatment. To determine incidence of complications related to nodal dissection are reduced with LVA.

Cancer-related lymphedema (CRLE) is a complex and lifelong implication of cancer treatment. Centres have reported rates of lymphedema following axillary node dissection of 39% (53% following adjuvant radiotherapy), and exceeding 73% following groin node dissection. Lymphedema can have significant quality of life (QoL) implications. Treatment, though helpful, is often burdensome, can require a second party to accomplish, and can be financially draining. Further, lymphedema is a chronic condition that cannot be eliminated once established. Many everyday activities, including self-care, employment, and social participation, as well as self-image, can be negatively impacted.

Given the high prevalence of CRLE, there is an urgency to investigate prophylaxis where possible. Prophylactic lymphaticovenous anastomosis offers this opportunity.

Although lymphaticovenous anastomosis (LVA) has been used for decades to treat existing lymphedema, more recently prophylactic LVA has been explored. Jørgensen et al's 2018 systematic review of 12 studies utilizing prophylactic LVA in cancer patients undergoing axilla or groin lymphadenectomy indicated a 2/3 reduction of CRLE in those treated prophylactically compared to those who did not receive prophylactic treatment.

More recently, Cakmakoglu et al reported on an immediate prophylactic approach whereby the LVA is performed at the time of nodal dissection utilizing fluorescing indocynanine green (ICG) and an operating microscope. This approach aided identification and assessment of the viability of lymphatic vessels in 96% of study cases, thereby augmenting the surgeon's ability to identify and choose the most appropriate vessels. Cakmakoglu's team performed the technique successfully on 22 patients. Of this 22, a single patient developed CRLE during the follow-up period (3 patients died of disease during the follow-up period but showed no sign of CRLE at their demise).

The outlook for LVA in combination with ICG looks promising but, to date, there has not been a Randomized Control Trial (RCT) on this prophylactic LVA technique. Thus, there is a need for robust RCTs utilizing a control group, having clearly defined outcome measures, investing in a significant follow-up period, and integrating blinded assessment in order to objectively demonstrate the impact of prophylactic LVA for patients.

Jørgensen et al's 2018 systematic review of prophylactic LVA case series and studies noted that, while the results were remarkable, the studies collected for the review did not have adequate control for bias and were quite heterogeneous in their cancer type, lymphadenectomy location, lymphedema classification, and assessment measures. QoL measures were not regularly integrated into assessment. Follow-up times varied from 6 months to 69 months with only 3 studies following for a minimum of 24 months.

Trial description:

Study participants will be comprised of patients undergoing lymphadenectomy for cutaneous malignancy. The participants will be block (axilla, groin) randomized using 2 equal groups (control/intervention) of 20 participants each. Participants assigned to the intervention arm will undergo prophylactic LVA as an addendum to their lymph node dissection. This will take place at time of lymphadenectomy surgery. Control participants will not have prophylactic LVA. Both groups will be blinded to treatment.

All participants will have limb volume measurements and photographs taken and the LYMQOL lymphedema-specific quality of life questionnaire administered at baseline (date of surgery) and at 6 month intervals for 24 months. Their recovery and surgical complications will be monitored as per the surgeon's usual followup schedule. At 24 months each participant will undergo a radionuclide lymphoscintigraphy to assess function and health of their lymphatic system. Unblinding will taken place at this juncture except in cases where necessary to unblind earlier to provide exceptional care.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons (>18 years of age) undergoing axilla or groin lymphadenectomy as part of cutaneous malignancy management.

Exclusion Criteria:

* Patients receiving a sentinel lymph node biopsy alone
* Patients with untreated in-transit disease on the upper or lower extremities
* Patients with established preoperative lymphedema
* Patients with post-thrombotic syndrome
* Pregnant patients
* Patients with a previous history of radiation therapy to the affected nodal basin or extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of lymphedema at 24 months post axillary or groin lymphadenectomy as assessed by limb volume over time. | 24 months
  Using a non-stretch measuring tape, circumferential measurements at 4cm intervals along the length of the contralateral limbs will be taken pre-surgery (baseline) and at 24 months. Limb volumes will be calculated. In the limb impacted by surgery, a 10% increase in volume from baseline to 24 months will be indicative of the development of lymphedema. In the case of significant weight gain or loss, comparison with the volume of the contralateral limb will also be used to evaluate presence of lymphedema in the surgical limb.
Quality of life impact as measured by LYMQOL PROM | 24 months
  A lymphedema quality of life patient reported outcome measure with specific arm and leg questionnaires called the LYMQOL will be used to measure quality of life. The scale uses a 4 point system for the majority of questions wherein a higher score indicates that lymphedema is having a greater negative impact on quality of life. A single final question uses a 10 point scale (poor to excellent) to rate one's quality of life overall with a higher score indicating greater quality of life. Comparison of quality of life scoring from baseline (pre-surgery) with scoring at 24 months post-surgery.

SECONDARY OUTCOMES:
Incidence of evidence of acute post-operative surgical complications | 24 months
  Diagnosis of complications such as cellulitis, dehiscence, lymphocele, and/or prolonged need for drain over 30days

CONTACTS AND LOCATIONS:
Overall Officials: Claire Temple-Oberle, MD, MSc, FRCSC, MMEd, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cakmakoglu C, Kwiecien GJ, Schwarz GS, Gastman B. Lymphaticovenous Bypass for Immediate Lymphatic Reconstruction in Locoregional Advanced Melanoma Patients. J Reconstr Microsurg. 2020 May;36(4):247-252. doi: 10.1055/s-0039-3401829. Epub 2019 Dec 31. PMID 31891946
- [Background] Rockson SG. Causes and consequences of lymphatic disease. Ann N Y Acad Sci. 2010 Oct;1207 Suppl 1:E2-6. doi: 10.1111/j.1749-6632.2010.05804.x. PMID 20961302
- [Background] Campanholi LL, Duprat JP, Fregnani JHTG. Incidence of le due to treating cutaneous melanoma. J Lymphoedema. 2011; 16(1): 30-34.
- [Background] Paskett ED, Dean JA, Oliveri JM, Harrop JP. Cancer-related lymphedema risk factors, diagnosis, treatment, and impact: a review. J Clin Oncol. 2012 Oct 20;30(30):3726-33. doi: 10.1200/JCO.2012.41.8574. Epub 2012 Sep 24. PMID 23008299
- [Background] Loprinzi PD, Cardinal BJ, Winters-Stone K, Smit E, Loprinzi CL. Physical activity and the risk of breast cancer recurrence: a literature review. Oncol Nurs Forum. 2012 May 1;39(3):269-74. doi: 10.1188/12.ONF.269-274. PMID 22543385
- [Background] Baibergenova A, Drucker AM, Shear NH. Hospitalizations for cellulitis in Canada: a database study. J Cutan Med Surg. 2014 Jan-Feb;18(1):33-7. doi: 10.2310/7750.2013.13075. PMID 24377471
- [Background] Tiwari P, Coriddi M, Salani R, Povoski SP. Breast and gynecologic cancer-related extremity lymphedema: a review of diagnostic modalities and management options. World J Surg Oncol. 2013 Sep 22;11:237. doi: 10.1186/1477-7819-11-237. PMID 24053624
- [Background] Dunberger G, Lindquist H, Waldenstrom AC, Nyberg T, Steineck G, Avall-Lundqvist E. Lower limb lymphedema in gynecological cancer survivors--effect on daily life functioning. Support Care Cancer. 2013 Nov;21(11):3063-70. doi: 10.1007/s00520-013-1879-3. Epub 2013 Jun 29. PMID 23812496
- [Background] Brayton KM, Hirsch AT, O Brien PJ, Cheville A, Karaca-Mandic P, Rockson SG. Lymphedema prevalence and treatment benefits in cancer: impact of a therapeutic intervention on health outcomes and costs. PLoS One. 2014 Dec 3;9(12):e114597. doi: 10.1371/journal.pone.0114597. eCollection 2014. PMID 25470383
- [Background] Gebruers N, Verbelen H, De Vrieze T, Coeck D, Tjalma W. Incidence and time path of lymphedema in sentinel node negative breast cancer patients: a systematic review. Arch Phys Med Rehabil. 2015 Jun;96(6):1131-9. doi: 10.1016/j.apmr.2015.01.014. Epub 2015 Jan 28. PMID 25637862
- [Background] Hormes JM, Bryan C, Lytle LA, Gross CR, Ahmed RL, Troxel AB, Schmitz KH. Impact of lymphedema and arm symptoms on quality of life in breast cancer survivors. Lymphology. 2010 Mar;43(1):1-13. PMID 20552814
- [Background] Jorgensen MG, Toyserkani NM, Sorensen JA. The effect of prophylactic lymphovenous anastomosis and shunts for preventing cancer-related lymphedema: a systematic review and meta-analysis. Microsurgery. 2018 Jul;38(5):576-585. doi: 10.1002/micr.30180. Epub 2017 Mar 28. PMID 28370317
- [Background] Garza RM, Chang DW. Lymphovenous bypass for the treatment of lymphedema. J Surg Oncol. 2018 Oct;118(5):743-749. doi: 10.1002/jso.25166. Epub 2018 Aug 11. PMID 30098298
- [Background] Hanson SE, Chang EI, Schaverien MV, Chu C, Selber JC, Hanasono MM. Controversies in Surgical Management of Lymphedema. Plast Reconstr Surg Glob Open. 2020 Mar 27;8(3):e2671. doi: 10.1097/GOX.0000000000002671. eCollection 2020 Mar. PMID 32537335
- [Derived] Jonsson EL, Fraser Hill WK, Saayman M, Yakaback S, Assadzadeh GE, Gregory McKinnon EJ, Temple-Oberle C. Pilot Study of Immediate Lymphatic Reconstruction (ILR) During Lymph Node Dissection for Node-Positive Melanoma: Feasibility, Safety, and Early Outcomes. J Surg Oncol. 2026 Jan;133(1):46-53. doi: 10.1002/jso.70127. Epub 2025 Nov 5. PMID 41190591
- [Derived] Temple-Oberle C, Nicholas C, Rojas-Garcia P. Current Controversies in Melanoma Treatment. Plast Reconstr Surg. 2023 Mar 1;151(3):495e-505e. doi: 10.1097/PRS.0000000000009936. Epub 2023 Feb 23. PMID 36821575
- [Derived] Deban M, Vallance P, Jost E, McKinnon JG, Temple-Oberle C. Higher Rate of Lymphedema with Inguinal versus Axillary Complete Lymph Node Dissection for Melanoma: A Potential Target for Immediate Lymphatic Reconstruction? Curr Oncol. 2022 Aug 11;29(8):5655-5663. doi: 10.3390/curroncol29080446. PMID 36005184